CLINICAL TRIAL: NCT02492256
Title: Atrial Ganglionated Plexi Ablation Guided by the SUMO Technology With and Without Conventional Pulmonary Vein Isolation in Persistent Atrial Fibrillation Patients: Prospective Randomized Study
Brief Title: Atrial Ganglionated Plexi Ablation Guided by the SUMO Technology With and Without Conventional Pulmonary Vein Isolation in Patients With Persistent AF
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPT15429
Record Dates: First submitted 2015-06-30; First posted 2015-07-08 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PVI group (Active Comparator): Conventional PVI by circumferential antral ablation according to standard procedures.
  Interventions: Device: Pulmonary vein isolation; Device: ILR implantation
- PVI+GP guided by SUMO technology group (Experimental): Conventional PVI by circumferential antral ablation according to standard procedures and atrial ganglionated plexi ablation guided by the SUMO technology.
  Interventions: Device: GP ablation guided by SUMO technology; Device: ILR implantation

INTERVENTIONS:
Device: Pulmonary vein isolation — CARTO- reconstruction LA, preferably during same rhythm as SUMO map (generally sinus rhythm) for use during registration of SUMO map in CARTO. Conventional PVI by circumferential antral ablation according to standard procedures. Exit and Entrance block conformation. Attempt to induce sustained atrial tachycardia. Optional mapping and ablation of post-ablation atrial tachycardia.
  Arms: PVI group
Device: GP ablation guided by SUMO technology — CARTO- reconstruction LA, preferably during same rhythm as SUMO map (generally sinus rhythm) for use during registration of SUMO map in CARTO. High frequency stimulation (HFS; 20-Hz frequency, 5-ms pulse duration, and 15-mA output) to access positive vagal response (the heart rate decreasing by 50% at baseline). RF Ablation of SUMO hotspots (in sinus rhythm if AF converts)
  • Target a region of 1.0-1.5 cm diameter around the SUMO 'hotspot'. Control HFS. Attempt to induce sustained atrial tachycardia. Optional mapping and ablation of post-ablation atrial tachycardia.
  Arms: PVI+GP guided by SUMO technology group
Device: ILR implantation — Implantation the ECG loop recorder according to standard procedure

SUMMARY:
Although circumferential pulmonary vein isolation (PVI) has been considered as the cornerstone for atrial fibrillation ablation, there has been a substantial recurrence rate. The investigators designed a prospectively randomized study to evaluate whether additional atrial ganglionated plexi ablation guided by the SUMO technology improves the clinical outcome in patients with persistent AF.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, age ≥ 18 and ≤ 80 years.
2. Persistent AF (ECG documentation).
3. Indication for AF ablation.
4. LVEF ≥ 50%
5. Able to provide written informed consent
6. Able to comply with the requirements of the study

Exclusion Criteria:

1. Reversible cause of atrial fibrillation
2. Previous AF ablation therapy
3. Clinical evidence of active coronary ischemia, significant valvular heart disease, or hemodynamically significant congenital cardiac abnormality
4. Recent (3 months) myocardial infarction (MI), stroke or transient ischemic attack (except if the patient had a DES implanted stent post-MI it would be one year)
5. Contra-indication to Iodine-123 Meta-iodobenzylguanidine (123I-mIBG), iodine, isoproterenol
6. Use of medication for non-cardiac medical conditions that is known to interfere with 123I-mIBG uptake and cannot be safely withheld for at least 24 hours prior to the D-SPECT study procedures
7. Inability to undergo D-SPECT and CT imaging

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-05 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Number of patients without AF/AFl/AT | 12 months

SECONDARY OUTCOMES:
Time to first recurrence of AF or atrial tachycardia (AF burden > 0,5%). | 12 month
Amount of mIBG uptake on 6 and 12 month DSPECT imaging in comparison to baseline D-SPECT. | 12 month

CONTACTS AND LOCATIONS:
Locations (1):
- State Research Institute of CIrculation Pathology Novosibirsk, Russian Federation, Novosibirsk, Russia